CLINICAL TRIAL: NCT04866758
Title: Improving Our Understanding of Suicidal Ideation in Cancer Survivors
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 17-7779.cc; P30CA046934 (NIH)
Record Dates: First submitted 2020-09-03; First posted 2021-04-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cancer Survivors: Ambulatory cancer population already seeking psychosocial support.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — All data gathered will be quantitative in nature. In addition to participant completed surveys, additional demographic, and diagnosis/treatment related information will be collected from the patient's electronic medical record via Health Data Compass. Subsequent data collected as part of the patient's standard psychosocial and cancer related care (i.e., health outcomes, future utilization of UCCC psychosocial services) will also be gathered. This subsequent data collection will not include further participation, but continued access to the patient's medical record. Protected health information collected for this project will include dates (e.g., birth dates, date of diagnosis, date since last treatment, death dates) and participant zip codes. No other identifiable data will be collected. A separate survey emailed to the participant at the end of the study will collect information regarding the participant's completion status of the survey.

SUMMARY:
The goal of this project is to assess the feasibility of collecting physiological and psychological data that will allow for preliminary investigation of predictors of suicidal ideation in an ambulatory cancer population already seeking psychosocial support.

DETAILED DESCRIPTION:
Exploratory analyses will be the first step to establishing possible predictive relationships. The long-term goal of this research is to identifying an integrated model of suicidal ideation in cancer, so that providers will be better able to identify appropriate screening methods to target patients at high risk for suicide. This information will ultimately inform the development of psychosocial interventions that specifically address the variables that increase suicide risk in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Be male or female, aged 18 or older.
4. Ambulatory oncology patients at the University of Colorado Cancer Center who are being provided psychosocial support services; specifically, having had at least one in-person meeting with a doctoral level clinical/counseling psychologist or masters level social worker.
5. Valid and private email account.

Exclusion Criteria:

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: An individual who fails to meet any of the inclusion criteria will be excluded from participation in this study. Mental health providers recruiting for this study may also use clinical judgment regarding appropriateness of participant for study (e.g., psychiatrically unstable).
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Suicidal Ideation Information | duration of study, no more than 2 weeks
  To evaluate the feasibility of data collection regarding physiological and psychological factors influencing suicidal ideation in cancer survivors

SECONDARY OUTCOMES:
Pain Intensity | duration of study, no more than 2 weeks
  The Brief Pain Inventory (BPI; Cleeland & Ryan, 1994) Pain Severity Scale consists of four 0-10 numerical rating scales evaluating (1) current pain as well as (2) worst (3) least and (4) average pain during the past 7 days. For this rating scale zero indicates, "no pain" while 10 indicates, "pain as bad as you can imagine". Averaging these four scores creates a composite score for pain severity. The measures has shown good internal consistency with Cronbach's alphas ranging from .78-.97 (Jensen, 2003).
Pain Interference | duration of study, no more than 2 weeks
  The BPI's Pain Interference Scale (Cleeland & Ryan, 1994) consists of seven items reflecting daily activities, including general activity, mood, walking ability, work, relationships, sleep, and enjoyment of life. A 0-10 numerical rating scale indicates the level of interference pain has had on each activity, with zero indicating, "does not interfere" and 10 indicating, "completely interferes". Averaging these seven scores creates a composite score for pain interference. The measure has shown good internal consistency with Cronbach's alphas ranging from .78-.91 (Jensen, 2003).
Symptom Burden/Severity | duration of study, no more than 2 weeks
  The MD Anderson Symptom Inventory (MDASI; Cleeland et al, 2000) is a self-report measure of cancer treatment-related symptoms. The measure includes 19 items, 13 of which comprise the symptom severity subscale and 6 of which comprise the symptom interference subscale. The symptom severity subscale asks patients to rate how severe various cancer-related symptoms (e.g., lack of appetite, dry mouth, fatigue) have been for them in the past 24 hours. Items on the symptom severity subscale are rated on a 0-10 numeric rating scale where 0 indicates "not present" and 10 indicates "as bad as you can imagine". The symptom interference subscale asks patients to rate the extent to which their symptoms have interfered with various domains of functioning (e.g. walking, enjoyment of life) in the past 24 hours. Items on the symptom interference subscale are rated on a 0-10 numeric rating scale where 0 indicates "did not interfere" and 10 indicates "interfered completely".
Physical Functioning | duration of study, no more than 2 weeks
  The PROMIS physical function short-form 6b (PF 6b) is a six item measure evaluating physical function using items from the National Institute of Health's Patient-Reported Outcomes Measurement Information System. Items on the PF 6b include questions such as "Does your health now limit you in doing two hours of physical labor?" and "Are you able to go up and down stairs at a normal pace?. Item responses are made on a 5-point Likert scale with one indicating "unable to do" and five indicating "without any difficulty". The measure has good internal reliability with a Cronbach's alpha of 0.94 (Jensen et al, 2015)
Health Related Quality of Life | duration of study, no more than 2 weeks
  The Functional Assessment of Cancer Therapy Scale-General (FACT-G; Cella et al, 1993) is a 27-item self-report measure of general cancer quality of life which includes physical, functional, social, and emotional well-being subscales. Items evaluate the endorsement of various cancer related symptoms, treatment related difficulties, or facets of psychosocial functioning within the past week. Item responses are rated on a 5-point Likert scale with zero indicating "not at all" and four indicating "very much". The measure has good internal reliability with a Cronbach's alpha of .89 (Cella et al, 1993).
Suicidal Ideation | duration of study, no more than 2 weeks
  The Suicidal Behaviors Questionnaire-Revised (SBQ-R; Osman et al, 2001) consists of four items which each tap into a different dimension of suicidality. Item 1 taps into lifetime suicidal ideation and/or suicide attempt. Item 2 assesses the frequency of suicidal ideation over the past twelve months. Item 3 assesses the threat of suicide attempt. Item 4 evaluates self-reported likelihood of suicidal behavior in the future. In adult general populations, this measure demonstrated 93% sensitivity and 95% specificity (Osman et al, 2001).
Experiential Avoidance | duration of study, no more than 2 weeks
  The Acceptance and Action Questionnaire-II (Bond et al, 2011) is a 7 item self-report measure assessing experiential avoidance. Item responses are rated on a seven-point Likert scale indicating the degree to which each statement is true for them ranging from (1) never true to (7) always true. The scale is scored by summing the seven items, with higher scores indicating lower levels of experiential acceptance. The measure has shown good internal reliability with a Cronbach's alpha of .84 (Bond et al, 2011).
Depression | duration of study, no more than 2 weeks
  The Patient Health Questionnaire (PHQ-9; Kroenke, Spitzer, & Williams, 2001) is a nine item self-report measure assessing the presence of DSM-IV criteria for major depressive episodes in the past two-week period. Item responses are rated on a four-point Likert scale with zero indicating "not at all" and three indicating "nearly every day". It has good internal reliability, with a Cronbach's alpha of 0.89 in primary care populations (Kroenke et al, 2001), and is endorsed by the American Society of Clinical Oncology (ASCO; Andersen et al, 2014) as a recommended screening tool for depression in cancer patients.
Hopelessness | duration of study, no more than 2 weeks
  The Hopelessness Assessment in Illness Questionnaire (Rosenfeld et al, 2011) is an eight item measure designed specifically to assess the construct of hopelessness as it pertains to terminally ill patients as it assesses hopelessness rather than awareness of prognosis. It is also shorter than other commonly used measures of hopelessness resulting in reduced patient burden. Each item has a three-choice anchored response format. The HAI has good internal reliability, with a Cronbach's alpha of 0.87. It demonstrated utility in predicting important psychosocial outcomes in terminally ill patients including suicidal ideation and desire for hastened death. It is recommended for use in other medically ill populations as well as terminally ill populations.
Anxiety | duration of study, no more than 2 weeks
  The GAD-7 (Spitzer, Kroenke, Williams & Lowe, 2006) is a seven-item self- report measure evaluating symptoms of anxiety associated with Generalized Anxiety Disorder experienced over the past two weeks. Items are rated on a 4-point Likert scale with zero indicating "not at all" and three indicating "nearly every day". It has good internal reliability, with a Cronbach's alpha of 0.92 (Spitzer et al. 2006), and is endorsed by ASCO as a recommended screening tool for anxiety in cancer patients (Andersen et al, 2014).
Demoralization | duration of study, no more than 2 weeks
  The Demoralization Scale-II (DS-II; Robinson et al., 2016a) is a sixteen-item scale that consists of two eight item subscales, meaning and purpose and distress and coping ability. A subtest analysis supported the use of a total score to estimate the construct of demoralization. Each item contains three response options (never, sometimes, and often). The DS-II has good internal consistence, as Cronbach's alpha for the total scale is .89. The scale demonstrated convergent validity with measures of quality of life and psychological distress in patients receiving palliative care (Robinson et al., 2016b).
Desire for Hastened Death | duration of study, no more than 2 weeks
  The Schedule of Attitudes Toward Hastened Death-Abbreviated (SAHD-A; Kolva, Rosenfeld, Liu, Pessin, Breitbart, 2016) is a six item measure self-report measure evaluating the desire for hastened death. The SAHD-A is short form of the Schedule of Attitudes toward Hastened Death (SAHD; Rosenfeld et al., 1999) the most commonly used self-report measure of desire for hastened death. The SAHD-A uses a True/False format and is comparable to the SAHD-A in its relationship to measures of psychological distress (i.e., depression, hopelessness, suicidal ideation), has good internal consistency (Cronbach's alpha = .83), and its short form reduces patient burden.

OTHER OUTCOMES:
Suicidality | 2 years
  Analyses will be stratified by cancer survivors with and without suicidal ideation. Descriptive statistics will be reported for clinical, demographic, and other study variables. Depending on data type and distribution, means, medians, or proportions will be reported with appropriate measures of data spread (i.e., standard deviation, range). Univariate analyses using the appropriate statistical tests (i.e., independent t-test, Wilcoxon rank sum, chi-square, logistic regression) will be performed to compare the two study groups. To allow for adjustment of potential confounders, multivariate analyses will be done using logistic regression techniques. Odds ratios and 95% confidence intervals will be reported. All tests will be two-sided and alpha will be set at 0.05. Data analyses and graphic results will be done using SAS (ver 9.4, SAS Institute, Cary, NC) and GraphPad Prism (ver 7.01, GraphPad Software Inc, La Jolla, CA).

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Studts, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No